CLINICAL TRIAL: NCT02188342
Title: Effectiveness of Short Term, High Intensity, Interval Exercise Training in Older Colorectal Cancer Patients in Improving Preoperative Fitness
Brief Title: Assessing The Effectiveness of a Preoperative High Intensity Interval Training Programme In Older Colorectal Cancer Patients
Acronym: HITCa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HITCa
Record Dates: First submitted 2014-07-10; First posted 2014-07-11 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Preoperative Care; Colorectal Neoplasms; Aged; Exercise
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIT exercise training (Experimental)
  Interventions: Behavioral: HIT

INTERVENTIONS:
Behavioral: HIT — 12 HIT exercise sessions in 31 days on a stationary cycle ergometer

SUMMARY:
The primary aim of this study is to determine whether an improvement in aerobic fitness, as judged by an increase in VO2peak, can be achieved within 31 days via HIT programme in a group of older, colorectal cancer patients.

DETAILED DESCRIPTION:
12 high intensity interval training exercise sessions on a static cycle ergometer, over a period of 31 days. Each session lasts 18 minutes.

At the beginning and end of the study the following measures will be used to assess change in fitness, body composition and muscle metabolism. DXA scan, USS of thigh, VO2 peak cycling test, short performance battery tests, quality of life questionnaires and muscle biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed colorectal cancer
* Offered curative treatment by the Royal Derby Hospital NHS Foundation Trust Colorectal Cancer Multidisciplinary Team
* Male and female
* 18-88 years of age

Exclusion Criteria:

* Uncontrolled hypertension (BP > 160/100),
* Angina,
* Heart failure (class III/IV),
* Cardiac arrthymias,
* Right to left cardiac shunt,
* Recent cardiac event,
* Previous stroke/TIA,
* Aneurysm (large vessel or intracranial),
* Severe respiratory disease including pulmonary hypertension,
* COPD/asthma with an FEV1 less than 1.5 l,
* Coagulation disorders,
* Scarring disorders.
* Current neoadjuvant chemo/radiotherapy
* Inability to complete the consent process Involvement in invasive research study in previous 3 months.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
VO2 peak | After 31 days of HIT
  Mean difference in VO2 peak following a HIT programme

SECONDARY OUTCOMES:
Anaerobic threshold | After 31 days of HIT
  Mean difference in anaerobic threshold following a HIT programme
Muscle protein synthesis | After 31 days of HIT
  Assessment of D2O evaluated muscle protein synthesis following HIT programme
Body composition | After 31 days of HIT
  DXA and USS assessed changes in lean muscle mass and architecture following a HIT programme
Feasibility | After 31 days of HIT
  Determination of patient compliance and adherence to HIT programme
Quality of life | After 31 days of HIT
  Quality of life and performance questionnaires to measure subjective outcomes (EQ-5D, IPAQ, DASI, WEMWBS)

CONTACTS AND LOCATIONS:
Overall Officials: John Williams, BSc MBChB FRCA PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Derby, Derbyshire, United Kingdom